CLINICAL TRIAL: NCT05215288
Title: Intermediate Size Expanded Access for the Use of ExoFlo in the Treatment of Abdominal Solid Organ Transplant Patients Who Are at Risk of Worsening Allograft Function With Conventional Immunosuppressive Therapy Alone
Brief Title: Expanded Access for Use of ExoFlo in Abdominal Solid Organ Transplant Patients
Status: No longer available | Type: Expanded Access
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DB-EF-TP_ASO-1a
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Solid Organ Transplant Rejection; Organ Rejection Transplants; Organ Rejection
Keywords: ExoFlo; Organ Rejection; Organ Rejection Transplants; Solid Organ Transplant Rejection

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: ExoFlo — Intravenous administration of bone marrow mesenchymal stem cell derived extracellular vesicles

SUMMARY:
This Expanded Access Protocol will provide access to the IMP ExoFlo for patients who have severe or life-threatening abdominal solid organ transplant rejection or who are evaluated and determined to be at high risk of progression to severe or life-threatening condition related to rejection of an abdominal solid organ transplant, at risk of worsening allograft function, or at risk of complications from current immunosuppressive therapeutic regimens.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this expanded access program is to evaluate safety and tolerability of ExoFlo in patients with graft inflammation, or worsening graft function, or evidence of rejection of an abdominal solid organ transplant despite conventional therapies. The secondary objective is to characterize the improvement seen in serum inflammatory markers and inflammation of solid abdominal organ.

Endpoints:

Primary Endpoint:

Incidence of AEs or SAEs.

Secondary Endpoint:

Improvement seen in serum inflammatory markers and inflammation of solid abdominal organ. This could include improvements seen in the following transplant types:

* Liver transplant: overall improved liver function, as seen by reduction in liver function test and improved albumin.
* Small bowel transplant: decreased inflammation on biopsy
* Pancreas: decreased amylase and lipase
* Multivisceral: any of the above criteria

Number of subjects: 20

Phase: Expanded Access Protocol

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, ages 18 to 75.
4. Previous abdominal solid organ transplant, including intestinal transplant.
5. Diagnosis of acute or chronic rejection / inflammation based on clinical observations, laboratory analysis, histological evaluation.
6. Diagnosis of worsening allograft function based on clinical observations, laboratory analysis, histological evaluation.
7. Failed primary and alternate standard of care therapies.
8. Serious or life-threatening condition or progressing to serious or life-threatening condition if not treated as evaluated by the treating physician.
9. In otherwise good general health as evidenced by medical history.
10. Male or female of reproductive potential must utilize a medically effective birth control method during from time of enrollment to 6 months after last dose of IMP.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Treatment with another investigational drug or other intervention within 30 days of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC
Locations (2):
- United States (2):
  - Direct Biologics Investigational Site, Palo Alto, California
  - Direct Biologics Investigational Site, San Francisco, California

REFERENCES:
- See also: Direct Biologics, LLC — https://directbiologics.com/